CLINICAL TRIAL: NCT03694808
Title: Non-inferiority Study of Adjuvanted vs. High Dose Flu Vaccine in Residents of Long Term Care
Brief Title: FLUAD vs. FLUZONE HD Influenza Vaccine in Residents of Long Term Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: David H. Canaday (Other)
Collaborators: Case Western Reserve University (Other); US Department of Veterans Affairs (U.S. Federal Agency); Brown University (Other); National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, David H. Canaday, Associate Professor of Medicine at Case Western Reserve University and Associate Director, Geriatric, Research, Education and Clinical Center at Louis Stokes Cleveland VA Medical Center, University Hospitals Cleveland Medical Center
Organization: University Hospitals Cleveland Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-27-29; 1R01AI129709-01A1 (NIH)
Record Dates: First submitted 2018-09-26; First posted 2018-10-03 (Actual); Results first posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Flu
Keywords: Flu; Vaccine
MeSH Terms: conditions — Influenza, Human | interventions — fluad vaccine

STUDY DESIGN:
Intervention Model Description: A non-inferiority randomized clinical trial to enroll 500 long term care (LTC) dwellers from at least one of 40 nursing homes sites in northern Ohio.
  Age 65 and older to receive either Fluad or HD vaccine at 1:1 ratio.
  Blood will be sampled pre- and post-vaccine and post-influenza season and coded for blinded laboratory analysis.
  Randomization by from randomizer.org software./RedCAP
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fluad Vaccine (Active Comparator): A single adjuvanted dose (AD) intramuscular injection
  Interventions: Drug: Fluad Vaccine
- Fluzone Vaccine (Active Comparator): A single high dose (HD) intramuscular injection
  Interventions: Drug: Fluzone HD Vaccine

INTERVENTIONS:
Drug: Fluad Vaccine — single adjuvanted dose (AD) intramuscular injection
  Arms: Fluad Vaccine
Drug: Fluzone HD Vaccine — single high dose (HD) intramuscular injection
  Arms: Fluzone Vaccine

SUMMARY:
Adjuvanted flu vaccine, Fluad, is not immunologically inferior to HD influenza vaccine in older persons living in long-term care.

DETAILED DESCRIPTION:
As the primary endpoint, this trial is be using pre- to post-vaccine changes in HAI titers to compare seroconversion rates and post-vaccination HAI titers to calculate the ratio of the geometric mean titers in the two treatment groups. HAI is an in vitro bioassay that determines a subject's serum levels of anti-influenza antibodies. The FDA uses this as a standard immunogenicity assay for licensure. The trial will follow guidelines set out in the FDA guidance document discussing non-inferiority immunogenicity studies. As additional methods to assess immunogenicity, an assessment of anti-NA by performing NA inhibition assays (NAI) and SVN assays will be added. A recent trial supported the use of NAI and SVN assays as a correlate for protection in a trial of geriatric subjects. A healthy human challenge model showed that NAI is more predictive of protection and reduced disease than HAI

In the large HD vaccine clinical efficacy trial (n=31,989) one third of subjects also had immunogenicity data that allowed looking for correlations of immune assays with protection. Their conclusions were that HAI and other immune assays are potential correlates of influenza vaccine protection in older adults, and that the protective thresholds for the HAI assay in the elderly appear consistent with those previously described for younger adults, provided the assay virus matches the circulating virus.

Significance Data compiled by CDC in 2011-2012 showed that there were 1,383,700 residents in NHs. Also about 4,742,500 patients received services from home health agencies, and 1,244,500 patients received services from hospices, collectively accounting for much of the frailest in the US. Overall, these provider sectors served over 8 million people annually (2013). This study will focus on residents in NHs but the findings of this study are highly relevant to persons frail enough to require such services in all of settings where the vast majority are at least 65 years old and thus appropriate for Fluad or HD, influenza vaccines licensed for this age group.

The SD influenza vaccine has diminished efficacy in the older population with the more debilitated LTC residents being among the worst responders yet with the highest mortality. Deaths due to pneumonia and influenza and chronic lung disease were 20 times higher among NH residents compared to community residents. The current availability of two vaccines specifically for the elderly that both appear to work better than SD vaccine begs the question: is the newer and less-costly Fluad vaccine non-inferior or even superior to HD vaccine? The proposed study aims to initially address non-inferiority using immunologic endpoints as this is feasible in the clinical trial R01 grant structure and a critical first step to obtain head-to-head data from the same trial, cohort and vaccine years. This proposed study itself may provide direct guidance on vaccine usage or inform a future trial assessing actual superiority should that be appropriate based on the results of this study.

HD vaccine is increasingly used by older Americans despite its greater cost over the SD vaccine and no preferential recommendation by the Advisory Committee on Immunization Practices (ACIP), the CDC committee responsible for making the vaccine recommendations for the U.S. A finding of non-inferiority in the primary endpoint would provide a strong rationale to consider using Fluad over HD that could result in some cost avoidance across large long-term care system in the U.S. The trial is not powered for a superiority analysis but in a non-inferiority trial if the findings are substantial enough they may show superiority.

In the normal seasonal setting, influenza strains drift antigenically and therefore vary from year to year. The CDC's prediction many months before the vaccination season sets the composition for the next season's vaccine, but does not always correctly anticipate the exact strain match that eventually actually circulates. There are Medicare claims data and modeling in the NH population that there is a significant increase in death and hospitalization in bad match over good match years particularly when A/H3N2 predominates. In those mismatched years in particular, heterologous immunity or immunity to other non-exact match strains becomes much more important if the vaccine is going to provide any benefit that season. Fluad is an adjuvanted vaccine that has been shown to have a more broad-based or heterologous immunity than SD vaccine that is not adjuvanted. HD is also not adjuvanted. Broad based immunity is especially desirable for A/H3N2 immunity as that has had 4 different circulating strains in the last 5 years while circulating A/H1N1 has been the same for 5 years; i.e., vaccine mismatch is more likely with the A/H3N2 circulating strain. A/H3N2 is associated with the majority of influenza hospitalizations and death among the elderly.

ELIGIBILITY:
Inclusion Criteria:

* > 65 years old
* Able to obtain consent from subject or legally authorized representative (subject to provide assent if cognitively/physically able to do so)
* Able to participate throughout the study period

Exclusion Criteria:

* Recent illness (within 30 days) severe enough to require hospitalization or physician-directed outpatient pharmacotherapy
* Administration of immunomodulatory agents (e.g. oral corticosteroids except prednisone < 10 mg daily, cyclosporine, and biologics (DMARDS) for Rheumatologic/Dermatologic conditions) in the last 3 months
* Cancer requiring treatment in the past three years, except for non- melanoma skin cancers or cancers that have clearly been cured or carry an excellent prognosis including prostate cancer.
* Myocardial infarction, major heart surgery (i.e. valve replacement or bypass surgery), stroke, deep vein thrombosis or pulmonary embolus in the past 4 months
* Allergies or history of significant adverse reactions to any component of influenza vaccine including egg protein and latex or after a previous dose of any influenza vaccine.
* History of Guillian-Barré Syndrome within 6 weeks of a prior influenza vaccine.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 478 (Actual)
Dates: Start 2018-09-23 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Canaday, MD, Principal Investigator — University Hospitals Cleveland Medical Center/Case Western Reserve University/Louis Stokes Cleveland VA Medical Center; Steven Gravenstein, MD, MPH, Principal Investigator — Brown University and Providence VA Medical Center
Locations (2):
- United States (2):
  - Louis Stokes Cleveland VA Medical Center, Cleveland, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ansaldi F, Bacilieri S, Durando P, Sticchi L, Valle L, Montomoli E, Icardi G, Gasparini R, Crovari P. Cross-protection by MF59-adjuvanted influenza vaccine: neutralizing and haemagglutination-inhibiting antibody activity against A(H3N2) drifted influenza viruses. Vaccine. 2008 Mar 17;26(12):1525-9. doi: 10.1016/j.vaccine.2008.01.019. Epub 2008 Feb 1. PMID 18294741
- [Background] Centers for Disease Control and Prevention (CDC). Estimates of deaths associated with seasonal influenza --- United States, 1976-2007. MMWR Morb Mortal Wkly Rep. 2010 Aug 27;59(33):1057-62. PMID 20798667
- [Background] DiazGranados CA, Dunning AJ, Kimmel M, Kirby D, Treanor J, Collins A, Pollak R, Christoff J, Earl J, Landolfi V, Martin E, Gurunathan S, Nathan R, Greenberg DP, Tornieporth NG, Decker MD, Talbot HK. Efficacy of high-dose versus standard-dose influenza vaccine in older adults. N Engl J Med. 2014 Aug 14;371(7):635-45. doi: 10.1056/NEJMoa1315727. PMID 25119609
- [Background] Dunning AJ, DiazGranados CA, Voloshen T, Hu B, Landolfi VA, Talbot HK. Correlates of Protection against Influenza in the Elderly: Results from an Influenza Vaccine Efficacy Trial. Clin Vaccine Immunol. 2016 Jan 13;23(3):228-35. doi: 10.1128/CVI.00604-15. PMID 26762363
- [Background] Falsey AR, Treanor JJ, Tornieporth N, Capellan J, Gorse GJ. Randomized, double-blind controlled phase 3 trial comparing the immunogenicity of high-dose and standard-dose influenza vaccine in adults 65 years of age and older. J Infect Dis. 2009 Jul 15;200(2):172-80. doi: 10.1086/599790. PMID 19508159
- [Background] Frey SE, Reyes MR, Reynales H, Bermal NN, Nicolay U, Narasimhan V, Forleo-Neto E, Arora AK. Comparison of the safety and immunogenicity of an MF59(R)-adjuvanted with a non-adjuvanted seasonal influenza vaccine in elderly subjects. Vaccine. 2014 Sep 3;32(39):5027-34. doi: 10.1016/j.vaccine.2014.07.013. Epub 2014 Jul 18. PMID 25045825
- [Background] Hancock K, Veguilla V, Lu X, Zhong W, Butler EN, Sun H, Liu F, Dong L, DeVos JR, Gargiullo PM, Brammer TL, Cox NJ, Tumpey TM, Katz JM. Cross-reactive antibody responses to the 2009 pandemic H1N1 influenza virus. N Engl J Med. 2009 Nov 12;361(20):1945-52. doi: 10.1056/NEJMoa0906453. Epub 2009 Sep 10. PMID 19745214
- [Background] Iob A, Brianti G, Zamparo E, Gallo T. Evidence of increased clinical protection of an MF59-adjuvant influenza vaccine compared to a non-adjuvant vaccine among elderly residents of long-term care facilities in Italy. Epidemiol Infect. 2005 Aug;133(4):687-93. doi: 10.1017/s0950268805003936. PMID 16050515
- [Background] Izurieta HS, Thadani N, Shay DK, Lu Y, Maurer A, Foppa IM, Franks R, Pratt D, Forshee RA, MaCurdy T, Worrall C, Howery AE, Kelman J. Comparative effectiveness of high-dose versus standard-dose influenza vaccines in US residents aged 65 years and older from 2012 to 2013 using Medicare data: a retrospective cohort analysis. Lancet Infect Dis. 2015 Mar;15(3):293-300. doi: 10.1016/S1473-3099(14)71087-4. Epub 2015 Feb 9. PMID 25672568
- [Background] Izurieta HS, Thadani N, Shay DK. Corrections. Comparative effectiveness of high-dose versus standard-dose influenza vaccines in US residents aged 65 years and older from 2012 to 2013 using Medicare data: a retrospective cohort analysis. Lancet Infect Dis. 2015 Mar;15(3):263. doi: 10.1016/S1473-3099(15)70070-8. No abstract available. PMID 25749223
- [Background] Mannino S, Villa M, Apolone G, Weiss NS, Groth N, Aquino I, Boldori L, Caramaschi F, Gattinoni A, Malchiodi G, Rothman KJ. Effectiveness of adjuvanted influenza vaccination in elderly subjects in northern Italy. Am J Epidemiol. 2012 Sep 15;176(6):527-33. doi: 10.1093/aje/kws313. Epub 2012 Aug 31. PMID 22940713
- [Background] Memoli MJ, Shaw PA, Han A, Czajkowski L, Reed S, Athota R, Bristol T, Fargis S, Risos K, Powers JH, Davey RT Jr, Taubenberger JK. Evaluation of Antihemagglutinin and Antineuraminidase Antibodies as Correlates of Protection in an Influenza A/H1N1 Virus Healthy Human Challenge Model. mBio. 2016 Apr 19;7(2):e00417-16. doi: 10.1128/mBio.00417-16. PMID 27094330
- [Background] Menec VH, MacWilliam L, Aoki FY. Hospitalizations and deaths due to respiratory illnesses during influenza seasons: a comparison of community residents, senior housing residents, and nursing home residents. J Gerontol A Biol Sci Med Sci. 2002 Oct;57(10):M629-35. doi: 10.1093/gerona/57.10.m629. PMID 12242314
- [Background] Pop-Vicas A, Rahman M, Gozalo PL, Gravenstein S, Mor V. Estimating the Effect of Influenza Vaccination on Nursing Home Residents' Morbidity and Mortality. J Am Geriatr Soc. 2015 Sep;63(9):1798-804. doi: 10.1111/jgs.13617. Epub 2015 Aug 17. PMID 26280675
- [Background] Richardson DM, Medvedeva EL, Roberts CB, Linkin DR; Centers for Disease Control and Prevention Epicenter Program. Comparative effectiveness of high-dose versus standard-dose influenza vaccination in community-dwelling veterans. Clin Infect Dis. 2015 Jul 15;61(2):171-6. doi: 10.1093/cid/civ261. Epub 2015 Mar 31. PMID 25829001
- [Background] Van Buynder PG, Konrad S, Van Buynder JL, Brodkin E, Krajden M, Ramler G, Bigham M. The comparative effectiveness of adjuvanted and unadjuvanted trivalent inactivated influenza vaccine (TIV) in the elderly. Vaccine. 2013 Dec 9;31(51):6122-8. doi: 10.1016/j.vaccine.2013.07.059. Epub 2013 Aug 6. PMID 23933368
- [Background] FDA. 2007. Guidance for Industry Clinical Data Needed to Support the Licensure of Seasonal Inactivated Influenza Vaccines. In Center for Biologics Evaluation and Research.
- [Background] 2013. Long-Term Care Services in the United States: 2013 Overview. In CDC, editor HHS, Disease Control and Prevention, National Center for Health Statistics, Hyattsville, Maryland.
- [Derived] Didion EM, Kass JD, Wilk DJ, Buss E, Frischmann SM, Rubeck S, Banks R, Wilson BM, Gravenstein S, Canaday DH. Which Enhanced Influenza Vaccine Has the Greatest Immunogenicity in Long-Term Care Residents: The Adjuvanted or the High-Dose Formulation? J Am Med Dir Assoc. 2025 Jul;26(7):105625. doi: 10.1016/j.jamda.2025.105625. Epub 2025 May 30. PMID 40373825

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 19 people were excluded prior to assignment to a group. People were excluded from the study if investigators failed to obtain all proper documentation on time (HIPPA, consent), if they withdrew consent, already got vaccine elsewhere, on antibiotics, ivermectin, refused vaccination, were hospitalized, left the facility prior to study completion for any reason.
Period: Overall Study
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Started | 240 | 219
Completed | 194 | 193
Not Completed | 46 | 26

BASELINE CHARACTERISTICS:
Population: 19 people were excluded prior to assignment. People were excluded from the study if investigators failed to obtain all proper documentation on time (HIPPA, consent), if they withdrew consent, already got vaccine elsewhere, on antibiotics, ivermectin, refused vaccination, were hospitalized, left the facility prior to study completion for any reason
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluad Vaccine | Fluzone Vaccine | Total
Number analyzed (Participants) | 194 | 193 | 387
Age, Continuous [Mean (Standard Deviation); unit: Years] | 79.5 (9.8) | 80.6 (9.3) | 80 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex was not reported on 2 people in the Fluad vaccine group.
  Participants
    number analyzed (Participants) | 192 | 193 | 385
    Female | 102 | 93 | 195
    Male | 90 | 100 | 190
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 183 | 181 | 364
  Unknown or Not Reported | 8 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 21 | 48
  White | 156 | 161 | 317
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Overall Hemagglutinin Inhibition (HAI) H1N1 Titer Between FLUAD and FLUZONE HD at 1 Month Post-vaccination.
Description: HAI is an in vitro bioassay testing subjects' sera for specific anti-influenza antibodies to each strain in the vaccine. Seroconversion is 4-fold rise in antibody titer. The FDA uses this as the standard immunogenicity assay for licensure. The investigators will follow the guidelines set out in the FDA guidance document on non-inferiority immunogenicity studies for the analysis plan.
Time Frame: 1 month post vaccine administration
Population: The total number analyzed represents the overall number of participants per group analyzed for both years combined. The total number analyzed per year is represented in the row value.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Number analyzed (Participants) | 192 | 190
Titer
  Year 1 (2018-2019): number analyzed (Participants) | 89 | 83
  Year 1 (2018-2019) | 213.4 [156.9 to 290.4] | 261.9 [192.3 to 356.6]
  Year 2 (2019-2020): number analyzed (Participants) | 103 | 107
  Year 2 (2019-2020) | 70.5 [53.5 to 92.9] | 67.2 [52.3 to 86.3]
Statistical Analysis 1: Comparison: Fluad Vaccine vs Fluzone Vaccine; Statistical Analysis for Year 1 (2018-2019); Test type: Non-Inferiority — Ratio of GMT (Fluzone/Fluad), upper bound of two-sided 95% CI should not exceed 1.5 for non-inferiority; t-test, 2 sided; ratio of GMT (Fluzone/Fluad) = 1.23, 95% CI 2-sided [0.8 to 1.89]
Statistical Analysis 2: Comparison: Fluad Vaccine vs Fluzone Vaccine; Statistical Analysis for Year 2 (2019-2020); Test type: Non-Inferiority — Ratio of GMT (Fluzone/Fluad), upper bound of two-sided 95% CI should not exceed 1.5 for non-inferiority; t-test, 2 sided; Ratio of GMT (Fluzone/Fluad) = 0.95, 95% CI 2-sided [0.66 to 1.38]

2. Primary Outcome: Overall Hemagglutinin Inhibition (HAI) H3N2 Titer Between FLUAD and FLUZONE HD at 1 Month Post-vaccination.
Description: as for outcome 1
Time Frame: 1 month post vaccine administration
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Number analyzed (Participants) | 194 | 193
Titer
  Year 1 (2018-2019): number analyzed (Participants) | 91 | 86
  Year 1 (2018-2019) | 375.5 [271.3 to 519.7] | 517.3 [380.8 to 702.6]
  Year 2 (2019-2020): number analyzed (Participants) | 103 | 107
  Year 2 (2019-2020) | 140.2 [96.9 to 202.7] | 120.4 [87.2 to 166.2]
Statistical Analysis 1: Comparison: Fluad Vaccine vs Fluzone Vaccine; Statistical Analysis for Year 1 (2018-2019); Test type: Non-Inferiority — Ratio of GMT (Fluzone/Fluad), upper bound of two-sided 95% CI should not exceed 1.5 for non-inferiority; t-test, 2 sided; Ratio of GMT (Fluzone/Fluad) = 1.38, 95% CI 2-sided [0.88 to 2.15]
Statistical Analysis 2: Comparison: Fluad Vaccine vs Fluzone Vaccine; Statistical Analysis for Year 2 (2019-2020); Test type: Non-Inferiority — Ratio of GMT (Fluzone/Fluad), upper bound of two-sided 95% CI should not exceed 1.5 for non-inferiority; t-test, 2 sided; Ratio of GMT (Fluzone/Fluad) = 0.86, 95% CI 2-sided [0.53 to 1.4]

3. Primary Outcome: Overall Hemagglutinin Inhibition (HAI) B Titer Between FLUAD and FLUZONE HD at 1 Month Post-vaccination.
Description: as for outcome 1
Time Frame: 1 month post vaccine administration
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Number analyzed (Participants) | 194 | 193
Titer
  Year 1 (2018-2019): number analyzed (Participants) | 91 | 86
  Year 1 (2018-2019) | 113.6 [87.6 to 146.8] | 210.4 [152.5 to 290.3]
  Year 2 (2019-2020): number analyzed (Participants) | 103 | 107
  Year 2 (2019-2020) | 75.5 [58.1 to 98.1] | 66.1 [51.1 to 85.5]
Statistical Analysis 1: Comparison: Fluad Vaccine vs Fluzone Vaccine; Statistical Analysis Year 1 (2018-2019); Test type: Non-Inferiority — Ratio of GMT (Fluzone/Fluad), upper bound of two-sided 95% CI should not exceed 1.5 for non-inferiority; t-test, 2 sided; Ratio of GMT (Fluzone/Fluad) = 1.85, 95% CI 2-sided [1.23 to 2.79]
Statistical Analysis 2: Comparison: Fluad Vaccine vs Fluzone Vaccine; Statistical Analysis Year 2 (2019-2020); Test type: Non-Inferiority — 2-sided t-test performed on log-transformed titers; estimate and 95% confidence interval of log-scale difference exponentiated to generate GMT ratio and its 95% CI below; t-test, 2 sided; Ratio of GMT (Fluzone/Fluad) = 0.88, 95% CI 2-sided [0.61 to 1.26]

4. Primary Outcome: Overall HAI H1N1 Seroconversion Rate Between FLUAD and FLUZONE HD at 1 Month Post-vaccination.
Description: as for outcome 1
Time Frame: 1 month post vaccine administration
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Number analyzed (Participants) | 192 | 190
percentage of participants
  Year 1 (2018-2019): number analyzed (Participants) | 89 | 83
  Year 1 (2018-2019) | 29.2 [20.3 to 40] | 44.6 [33.8 to 55.9]
  Year 2 (2019-2020): number analyzed (Participants) | 103 | 107
  Year 2 (2019-2020) | 48.5 [38.7 to 58.5] | 43 [33.6 to 52.9]
Statistical Analysis 1: Comparison: Fluad Vaccine vs Fluzone Vaccine; Statistical Analysis Year 1 (2018-2019); Test type: Non-Inferiority — Difference between seroconversion rates (Fluzone - Fluad), upper bound of two-sided 95% CI of difference should not exceed 10 percentage points for non-inferiority; Test of proportions; 2sided proportions test to estimate 95% CI difference in seroconversion rates; upper limit differences compared to 10%, per non-inferiority guidance; Difference in proportions = 0.154, 95% CI 2-sided [-0.001 to 0.308]
Statistical Analysis 2: Comparison: Fluad Vaccine vs Fluzone Vaccine; Statistical Analysis Year 2 (2019-2020); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Test of proportions; [statistical method as in outcome 4, analysis 1]; Difference in proportions = -0.056, 95% CI 2-sided [-0.2 to 0.089]

5. Primary Outcome: Overall HAI H3N2 Seroconversion Rate Between FLUAD and FLUZONE HD at 1 Month Post-vaccination.
Description: as for outcome 1
Time Frame: 1 month post vaccine administration
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Number analyzed (Participants) | 194 | 193
percentage of participants
  Year 1 (2018-2019): number analyzed (Participants) | 91 | 86
  Year 1 (2018-2019) | 35.2 [25.6 to 46] | 57 [45.9 to 67.5]
  Year 2 (2019-2020): number analyzed (Participants) | 103 | 107
  Year 2 (2019-2020) | 70.9 [61 to 79.2] | 70.1 [60.4 to 78.4]
Statistical Analysis 1: Comparison: Fluad Vaccine vs Fluzone Vaccine; Statistical Analysis Year 1 (2018-2019); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Test of proportions; [statistical method as in outcome 4, analysis 1]; Difference in proportions = 0.218, 95% CI 2-sided [0.063 to 0.373]
Statistical Analysis 2: Comparison: Fluad Vaccine vs Fluzone Vaccine; Statistical Analysis Year 2 (2019-2020); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Test of proportions; [statistical method as in outcome 4, analysis 1]; Difference in proportions = -0.008, 95% CI 2-sided [-0.139 to 0.123]

6. Primary Outcome: Overall HAI B Seroconversion Rate Between FLUAD and FLUZONE HD at 1 Month Post-vaccination.
Description: as for outcome 1
Time Frame: 1 month post vaccine administration
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Number analyzed (Participants) | 194 | 193
percentage of participants
  Year 1 (2018-2019): number analyzed (Participants) | 91 | 86
  Year 1 (2018-2019) | 34.1 [24.7 to 44.8] | 47.7 [36.9 to 58.7]
  Year 2 (2019-2020): number analyzed (Participants) | 103 | 107
  Year 2 (2019-2020) | 36.9 [27.8 to 47] | 39.3 [30.1 to 49.2]
Statistical Analysis 1: Comparison: Fluad Vaccine vs Fluzone Vaccine; Statistical Analysis Year 1 (2018-2019); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Test of proportions; [statistical method as in outcome 4, analysis 1]; Difference in proportions = 0.136, 95% CI 2-sided [-0.019 to 0.291]
Statistical Analysis 2: Comparison: Fluad Vaccine vs Fluzone Vaccine; Statistical Analysis Year 2 (2019-2020); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Test of proportions; [statistical method as in outcome 4, analysis 1]; Difference in proportions = 0.024, 95% CI 2-sided [-0.117 to 0.164]

7. Secondary Outcome: Overall Neuraminidase Inhibition (NAI) H1N1 Titer Between FLUAD and FLUZONE HD at 1 Month Post-vaccination.
Description: Neuraminidase inhibition (NAI) assays will be performed to measure anti-neuraminidase titers. Seroconversion is 4-fold rise in antibody titer.
Time Frame: 1 month post vaccine administration
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Number analyzed (Participants) | 192 | 189
Titer
  Year 1 (2018-2019): number analyzed (Participants) | 89 | 83
  Year 1 (2018-2019) | 167.7 [128.2 to 219.3] | 71.8 [53 to 97.3]
  Year 2 (2019-2020): number analyzed (Participants) | 103 | 106
  Year 2 (2019-2020) | 666.4 [497.7 to 892.3] | 297.8 [214.3 to 413.8]
Statistical Analysis 1: Comparison: Fluad Vaccine vs Fluzone Vaccine; Statistical Analysis Year 1 (2018-2019); Test type: Non-Inferiority — Ratio of GMT (Fluzone/Fluad), upper bound of two-sided 95% CI should not exceed 1.5 for non-inferiority; t-test, 2 sided; Ratio of GMT (Fluzone/Fluad) = 0.43, 95% CI 2-sided [0.29 to 0.64]
Statistical Analysis 2: Comparison: Fluad Vaccine vs Fluzone Vaccine; Statistical Analysis Year 2 (2019-2020); Test type: Non-Inferiority — Ratio of GMT (Fluzone/Fluad), upper bound of two-sided 95% CI should not exceed 1.5 for non-inferiority; t-test, 2 sided; Ratio of GMT (Fluzone/Fluad) = 0.45, 95% CI 2-sided [0.29 to 0.69]

8. Secondary Outcome: Overall Neuraminidase Inhibition (NAI) H3N2 Titer Between FLUAD and FLUZONE HD at 1 Month Post-vaccination.
Description: as for outcome 7
Time Frame: 1 month post vaccine administration
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Number analyzed (Participants) | 194 | 192
Titer
  Year 1 (2018-2019): number analyzed (Participants) | 91 | 86
  Year 1 (2018-2019) | 27.3 [23.3 to 32.1] | 24.9 [20.6 to 30.1]
  Year 2 (2019-2020): number analyzed (Participants) | 103 | 106
  Year 2 (2019-2020) | 46.7 [37.1 to 58.8] | 44.7 [35.4 to 56.4]
Statistical Analysis 1: Comparison: Fluad Vaccine vs Fluzone Vaccine; Statistical Analysis Year 1 (2018-2019); Test type: Non-Inferiority — Ratio of GMT (Fluzone/Fluad), upper bound of two-sided 95% CI should not exceed 1.5 for non-inferiority; t-test, 2 sided; Ratio of GMT (Fluzone/Fluad) = 0.91, 95% CI 2-sided [0.71 to 1.16]
Statistical Analysis 2: Comparison: Fluad Vaccine vs Fluzone Vaccine; Statistical Analysis Year 2 (2019-2020); Test type: Non-Inferiority — Ratio of GMT (Fluzone/Fluad), upper bound of two-sided 95% CI should not exceed 1.5 for non-inferiority; t-test, 2 sided; Ratio of GMT (Fluzone/Fluad) = 0.96, 95% CI 2-sided [0.69 to 1.33]

9. Secondary Outcome: Overall H1N1 NAI Seroconversion Rate Between FLUAD and FLUZONE HD at 1 Month Post-vaccination.
Description: as for outcome 7
Time Frame: 1 month post vaccine administration
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Number analyzed (Participants) | 192 | 189
percentage of participants
  Year 1 (2018-2019): number analyzed (Participants) | 89 | 83
  Year 1 (2018-2019) | 64 [53.1 to 73.7] | 9.6 [4.6 to 18.6]
  Year 2 (2019-2020): number analyzed (Participants) | 103 | 106
  Year 2 (2019-2020) | 60.2 [50.1 to 69.6] | 43.4 [33.9 to 53.4]
Statistical Analysis 1: Comparison: Fluad Vaccine vs Fluzone Vaccine; Statistical Analysis Year 1 (2018-2019); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Test of proportions; [statistical method as in outcome 4, analysis 1]; Difference in proportions = -0.544, 95% CI 2-sided [-0.674 to -0.414]
Statistical Analysis 2: Comparison: Fluad Vaccine vs Fluzone Vaccine; Statistical Analysis Year 2 (2019-2020); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Test of proportions; [statistical method as in outcome 4, analysis 1]; Difference in proportions = -0.168, 95% CI 2-sided [-0.311 to -0.025]

10. Secondary Outcome: Overall NAI H3N2 Seroconversion Rate Between FLUAD and FLUZONE HD at 1 Month Post-vaccination.
Description: as for outcome 7
Time Frame: 1 month post vaccine administration
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Number analyzed (Participants) | 194 | 192
percentage of participants
  Year 1 (2018-2019): number analyzed (Participants) | 91 | 86
  Year 1 (2018-2019) | 20.9 [13.3 to 30.9] | 10.5 [5.2 to 19.4]
  Year 2 (2019-2020): number analyzed (Participants) | 103 | 106
  Year 2 (2019-2020) | 32 [23.4 to 42.1] | 20.8 [13.7 to 29.9]
Statistical Analysis 1: Comparison: Fluad Vaccine vs Fluzone Vaccine; Statistical Analysis Year 1 (2018-2019); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Test of proportions; [statistical method as in outcome 4, analysis 1]; Difference in proportions = -0.104, 95% CI 2-sided [-0.221 to 0.013]
Statistical Analysis 2: Comparison: Fluad Vaccine vs Fluzone Vaccine; Statistical Analysis Year 2 (2019-2020); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Test of proportions; [statistical method as in outcome 4, analysis 1]; Difference of proportions = -0.113, 95% CI 2-sided [-0.241 to 0.015]

11. Secondary Outcome: Overall Serum Virus Neutralization (SVN) H1N1 Titer Between FLUAD and FLUZONE HD at 1 Month Post-vaccination.
Description: Serum virus neutralization (SVN) assays will be performed to measure the ability of serum to inhibit influenza infection.
Time Frame: 1 month post vaccine administration
Population: SVN assay was only performed on samples for the 2018-2019 flu season. The 2019-2020 assays were not performed due to interruption by SARS-Cov-2 pandemic.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Number analyzed (Participants) | 65 | 67
Titer | 675.7 [532.2 to 872.7] | 791.3 [647.7 to 966.7]

12. Secondary Outcome: Heterologous Immunity at 1 Month Post-vaccination Will be Compared Between FLUAD and FLUZONE HD.
Description: Hemagglutinin inhibition (HAI), neuraminidase inhibition (NAI) assays and serum virus neutralization (SVN) assays will be performed with heterologous A/H3N2 strains to determine if Fluad has an increased breadth of both B and T cell responses as would be predicted from an adjuvanted vaccine.
Time Frame: 1 month post vaccine administration
Population: No data was collected
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Number analyzed (Participants) | 0 | 0

13. Other Pre Specified Outcome: To Pilot Clinical Objective: Efficacy of FLUAD Will be Compared to FLUZONE HD.
Description: A record review and a blood 2 weeks after the influenza season is over will be done. From a record review the dates and diagnoses of hospitalizations and/or "influenza like illness" (ILI) will be recorded. Serologic evidence of influenza infection ( >=4-fold titer rise beyond the post-vaccine titers) will be determined from the remote blood draw. An exploratory analysis will be performed comparing the efficacy of the two vaccines.
Time Frame: 6-8 months post vaccine administration
Population: No data collected
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Overall Serum Virus Neutralization (SVN) H3N2 Titer Between FLUAD and FLUZONE HD at 1 Month Post-vaccination.
Description: as for outcome 11
Time Frame: 1 month post vaccine administration
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Number analyzed (Participants) | 66 | 65
Titer | 270.8 [180 to 407.3] | 405.0 [279.9 to 586]

15. Secondary Outcome: Overall Serum Virus Neutralization (SVN) H1N1 Seroconversion Between FLUAD and FLUZONE HD at 1 Month Post-vaccination.
Description: as for outcome 11
Time Frame: 1 month post vaccine administration
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Number analyzed (Participants) | 65 | 67
percentage of participants | 32.3 [21.5 to 45.2] | 31.3 [20.9 to 44]

16. Secondary Outcome: Overall Serum Virus Neutralization (SVN) H3N2 Seroconversion Between FLUAD and FLUZONE HD at 1 Month Post-vaccination.
Description: as for outcome 11
Time Frame: 1 month post vaccine administration
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fluad Vaccine | Fluzone Vaccine
Number analyzed (Participants) | 66 | 65
percentage of participants | 21.2 [12.5 to 33.3] | 43.1 [31.1 to 55.9]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was only monitored/assessed two weeks following the final blood draw (up to 8 months post vaccine administration). Serious and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: All-Cause Mortality was only monitored/assessed two weeks following the final blood draw (up to 8 months post vaccine administration). Serious and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Fluad Vaccine | Fluzone Vaccine
All-Cause Mortality (participants affected / at risk) | 1/194 | 1/193
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
1. For all SVN related outcomes (11, 13, 14, 15) data was only collected for the 2018-2019 season
2. >38% of values are at upper limit of detection (25% of Day 0 and >50% of Day 28 values)

Thus, the assay fails to capture any variability in values > 1000. Given how many subjects have values in this range, we are unable to accurately summarize group differences; and a seroconversion endpoint that requires measuring change from d0 to d28 cannot be validly measured given this limitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/08/NCT03694808/Prot_SAP_000.pdf